CLINICAL TRIAL: NCT00001173
Title: Studies of In Vitro B Lymphocyte Responses in Subjects Receiving Tetanus Toxoid Booster Immunization
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 800070; 80-I-0070
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-06

CONDITIONS: Healthy
Keywords: B Cells; Humoral Immunity; Lymphocytes; Tetanus Toxoid
MeSH Terms: conditions — Tetanus

SUMMARY:
One of the major interests of this laboratory is the characterization of the cellular subpopulations involved in the triggering and immunoregulation of B lymphocytes to produce antibodies. We are assessing the responses of individuals to produce antibodies against newly encountered antigens such as keyhole limpet hemocyanin (KLH) (approved project number 77-I-0130) and propose to assess the amnestic responses to the previously encountered antigen, tetanus toxoid. The purpose of this protocol is to add this recall antigen to our repertoire of antigens used to evaluate the immune response in man.

Booster immunization with tetanus/diphtheria toxoid has now been used for several years by a number of clinical immunology laboratories throughout the country to assess B cell related immunologic profiles in patients and control normal subjects. We have recently developed a sensitive ELISA assay for IgM and IgG in vitro specific antibody responses against tetanus toxoid. This will allow us to carefully and precisely monitor the evolution and immunoregulation of the human B cell responses to this recall antigen. This is of particular importance and relevance to us in our ongoing studies of a number of diseases characterized by abnormalities of immunologic reactivity, including those treated with various regimens of immunosuppressive agents.

DETAILED DESCRIPTION:
One of the major interests of this laboratory is the characterization of the cellular subpopulations involved in the triggering and immunoregulation of B lymphocytes to produce antibodies. We are assessing the responses of individuals to produce antibodies against newly encountered antigens such as keyhole limpet hemocyanin (KLH) (approved project number 77-I-0130) and propose to assess the amnestic responses to the previously encountered antigen, tetanus toxoid. The purpose of this protocol is to add this recall antigen to our repertoire of antigens used to evaluate the immune response in man.

Booster immunization with tetanus/diphtheria toxoid has now been used for several years by a number of clinical immunology laboratories throughout the country to assess B cell related immunologic profiles in patients and control normal subjects. We have recently developed a sensitive ELISA assay for IgM and IgG in vitro specific antibody responses against tetanus toxoid. This will allow us to carefully and precisely monitor the evolution and immunoregulation of the human B cell responses to this recall antigen. This is of particular importance and relevance to us in our ongoing studies of a number of diseases characterized by abnormalities of immunologic reactivity, including those treated with various regimens of immunosuppressive agents.

ELIGIBILITY:
Male and female patients 18 years and older.

Patients admitted to the Clinical Center under other approved research protocols designed to investigate immune mediated or inflammatory diseases and who have not been immunized to tetanus toxoid within 6 months.

No pregnant women.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200
Dates: Start 1980-06; Study Completion 2000-06

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Allergy and Infectious Diseases (NIAID), Bethesda, Maryland, United States